CLINICAL TRIAL: NCT01325142
Title: Genetic Risk of Osteonecrosis of the Jaw (ONJ) in Patients With Metastatic Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Indiana University (Other); M.D. Anderson Cancer Center (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Catherine Van Poznak, Priniciple Investigator, University of Michigan
Other Study IDs: HUM00040101; 5K23DE020197-02 (NIH)
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Bone Diseases; Metastases; Osteonecrosis; Bisphosphonate-Associated Osteonecrosis of the Jaw
Keywords: Osteonecrosis of the Jaw (ONJ)
MeSH Terms: conditions — Bone Diseases; Neoplasm Metastasis; Osteonecrosis; Bisphosphonate-Associated Osteonecrosis of the Jaw

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — paraffin embedded tissue block and/or WBC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ONJ: Patient with cancer involving the bone treated with osteoclast inhibitor (bisphosphonate) and has developed ONJ
- No ONJ: Patient with cancer involving the bone treated with osteoclast inhibitor (bisphosphonate) and has NOT developed ONJ

SUMMARY:
This study seeks to identify risk factors associated with the development of a jaw condition seen in patients with cancer treated with certain medications.

DETAILED DESCRIPTION:
The goal of this research is to build an index of risk for estimating an individual's risk of developing osteonecrosis of the jaw (ONJ). The bisphosphonates are an important supportive therapy in the care of patients with metastatic bone disease; they are able to prevent catastrophic events such as fracture and spinal cord compression. However, ONJ has been associated with the use of the bisphosphonates and ONJ carries significant morbidity. Presently, there are insufficient data to calculate the ONJ risk benefit ratio of bisphosphonate use. An ONJ risk assessment tool would improve both the oncologist's and the dental health professional the ability to anticipate and potentially mitigate oral toxicities from bisphosphonate therapy.

This protocol consists of a case (ONJ) control (no ONJ) study to identify factors associated with the risk of ONJ and to build an index predictive of an individual's risk of developing ONJ. The index of ONJ risk will be comprised of clinical, epidemiologic and genetic factors

ELIGIBILITY:
Inclusion Criteria:

* The study candidate must have sufficient Formalin Fixed Paraffin Embedded (FFPE)Specimens (lymph node or tumor) for DNA extraction available for study SNP assessment
* Patients over the age of 21 with a histologically confirmed diagnosis of cancer who have received nitrogen containing bisphosphonate therapy for metastatic bone disease.
* FFPE tissues are to have been removed for clinical indication and sufficience study volume of specimen must be available in an established tissue repository.
* - Study FFPE tissues include:

  * formalin fixed paraffin embedded leukocytes from lymph nodes with or without involvement by tumor AND/OR
  * formalin fixed paraffin embedded tumor tissue (tumor block without invasive cancer is acceptable if the specimen is believed to be sufficiently cellular (breast tissue or noninvasive cancer) to yield adequate DNA)
* Medical records available for data abstraction

Exclusion Criteria:

* Insufficient specimen available to perform the assays proposed for specimen DNA analysis
* No accessable medical records

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Academic medical center(s)
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To identify clinical and epidemiologic characteristics associated with ONJ in patients with metastatic bone disease treated with a nitrogen containing bisphosphonate. | 2009-2014
  analysis is ongoing
To identify single nucleotide polymorphisms (SNPs) in genes affected by osteoclast inhibiting therapy that are associated with an increased risk of developing ONJ in patients with metastatic bone disease treated with nitrogen containing bisphosphonates. | 2009-2014
  analysis is ongoing
To generate a multifactorial index of ONJ risk by multivariate analysis of the clinical, epidemiologic and genetic factors | 2009-2014
  analysis is ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Van Poznak, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States